CLINICAL TRIAL: NCT06032208
Title: An Extension of an Interventional Study to Assess the Effect of Expanded Dialysis (HDx-Theranova) on Patient Reported Symptoms Using London Evaluation of Illness (LEVIL)
Brief Title: An Extension to Assess the Effect of Expanded Dialysis on Patient Reported Symptoms Using LEVIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Chris McIntyre, Professor of Medicine, Medical Biophysics and Paediatrics, Robert Lindsay Chair of Dialysis Research and Innovation, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 123850
Record Dates: First submitted 2023-08-31; First posted 2023-09-11 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Large middle molecules; Theranova
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Study visits take place within the patients usual hemodialysis unit consistent with their routinely scheduled dialysis sessions. Beginning week 5 participants will use the Theranova dialyzer until the end of dialysis week 28. Participants will answer 9 questions at least (1-3 times weekly) - weeks 1 through 28 (entire length of study) using the LEVIL application.
  Furthermore, participants answer a single Time-to-Recovery question between weeks 1-4 and repeated at week 28 to get more information on recovery time after dialysis in addition to completing Creyos (cognitive testing formally Cambridge Brain Sciences), as well as Sexual Desire Inventory-2 testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receiving Hemodialysis (Experimental): A group of hemodialysis patients will be receiving the Theranova dialyzer during their regular scheduled dialysis sessions to remove larger middle molecules.
  Interventions: Device: Theranova Dialyzer

INTERVENTIONS:
Device: Theranova Dialyzer — The Theranova dialyzer will be used for each of the hemodialysis treatments beginning week 5 and ending at the end of dialysis week 28. This will allow us to compare patient reported symptoms in weeks 1-4 on their usual dialyzer with with their symptoms on the Theranova dialyzer.

SUMMARY:
Investigators know that many patients who are on dialysis suffer from burden of unwanted symptoms, which can affect quality of life. The understanding and treatment of symptom burden by healthcare providers is limited and should be recognized as a high priority in the care of the dialysis population. In this study, the investigators will be assessing symptom burden using the London Evaluation of Illness "LEVIL," an application based platform where patients self-report their symptoms with one to three hemodialysis treatments per week for 28 weeks. The investigators would like to compare the currently available dialyzer with a new dialyzer that is capable of removing solutes of higher molecular weight that may or may not cause patients to experience symptoms related to increased amounts of toxins in their blood.

DETAILED DESCRIPTION:
Baxter Canada has an expanded hemodialysis (HDx) membrane called the "Theranova", which is capable of removing solutes of higher molecular weight. Although this clearly has biochemical advantages it is not known at this time if the removal of larger middle molecules can have a direct and immediate effect on patients reported symptoms and quality of life. In short, do people actually feel better?

Given the way many quality of life measurements fluctuate around the dialysis week, the investigators propose to utilize a dynamic tool. The investigators will be assessing symptom burden using the London Evaluation of Illness "LEVIL" an application based platform where patients self-report their symptoms with at least one hemodialysis treatment. Reports are generated immediately and in real-time, which cannot be accomplished with other symptom management tools. This allows the investigators to track study changes and benchmark observations to previously established baseline values. The investigators are excited to see if there is an imminent effect on how patients feel using the Theranova dialyzer.

The study is investigator initiated and the principal investigator has secured modest funding from Baxter to allow support for the core study team and the introduction and maintenance of the LEVIL evaluation platform at other centers. Baxter have also provided some dialyzer support and will work with individual centers to ensure that there is no consumable increment of cost associated with participation.

The study is 28 weeks in length:

* LEVIL entries with at least 1 to 3 hemodialysis treatments each week for 28 weeks.
* Implementation of Theranova dialyzer from week 5 until the end of week 28.
* Creyos (cognitive testing) one time at baseline (between weeks 1 to 4) and again during week 28.
* Sexual Desire questionnaire one time at baseline (between weeks 1 to 4) and again during week 28.

ELIGIBILITY:
Inclusion Criteria:

* Conventional thrice weekly HD schedule
* Must be on chronic hemodialysis for at least 3 months
* Age ≥18 years
* Willing and able to give informed consent

Exclusion Criteria:

* Active infection (may enroll once infection is cleared)
* Patients receiving daily hemodialysis treatment
* Patients currently receiving Hemodiafiltration (HDF), Hemofiltration (HF) or Isolated ultrafiltration (ISO UF) more than once in three months
* Visual impairment
* History of neurocognitive impairment
* History of stroke (CVA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine if the clearance of larger middle molecular weight toxins using medium-cut-off dialyzer (HDx -Theranova) effects patient reported symptoms as determined by LEVIL. | Beginning week 1 and ending at the end of dialysis on week 28.
  The primary outcome will be a change (from patient's own baseline) in general well-being, pain, sleep. breathing, energy, appetite, itch, restless legs, and recovery from hemodialysis when using the Theranova dialyzer. These parameters will be measured using the LEVIL, an electronic application based visual analog scale.
  The scale indicates Very Poor on the left and Excellent to the right or Extreme on the left to No Problem on the right. Participants will use their finger and slide the scale to indicate which best describes how they feel.

SECONDARY OUTCOMES:
Determine if the clearance of larger middle molecular weight toxins using medium-cut-off dialyzer (HDx-Theranova) effects cognition. | Between weeks 1 & 4 and repeated during week 28
  Cognitive Testing measured using Creyos (formally Cambridge Brain Sciences) web-based application at baseline (between weeks 1 & 4) and repeated at week 28.
  Creyos consists of tasks that are separated into domains of reasoning, short term memory, and verbal abilities:
  1. Odd one Out (patterns), 2. Digit Span (number sequence), 3. Paired Association Task, 5. Rotations Task, 6. Monkey Ladder Task
Determine if the clearance of larger middle molecular weight toxins using medium-cut-off dialyzer (HDx-Theranova) effects sexual desire | Between weeks 1 & 4 and repeated during week 28
  Parameters will be measured using Sexual Desires Inventory-2 (SDI-2) an anonymous web-based platform at baseline (between weeks 1 & 4) and repeated at week 28.
  SDI-2 is a multiple choice platform where participants will privately answer questions that best describes how they feel. (eg. not at all, once a month, once every two months, once a week, twice a week, 3 to 4 times a week, once a day, more then once a day) A score will be populated within the app and the score will be recorded only.
Determine if the clearance of larger middle molecular weight toxins using medium-cut-off dialyzer (HDx-Theranova) effects dialysis recovery time compared to high-flux dialysis membrane. | Between weeks 1 & 4 and repeated during week 28
  Parameters will be measured using Time-to-Recovery question at baseline (between weeks 1 & 4) and repeated at week 28.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McIntyre, MBBS DM, Principal Investigator — London Heath Sciences Centre
Locations (2):
- Canada (2):
  - Victoria Hospital, London Health Sciences Centre, London, Ontario
  - Westmount Kidney Care Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No